CLINICAL TRIAL: NCT04126499
Title: Observational Retrospective Study to Characterise Patients Receiving Benralizumab in the Framework of an Individualized Access Program in Spain
Brief Title: Study to Characterise Patients Receiving Benralizumab in the Framework of an Individualized Access Program in Spain
Acronym: ORBE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00052
Record Dates: First submitted 2019-09-25; First posted 2019-10-15 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Severe Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

SUMMARY:
Observational, retrospective study in adults (≥18 years) with severe asthma (maintenance treatment with high dose inhaled corticosteroids combined with long-acting agonist β2) and eosinophilic phenotype, who at the discretion of the investigator were candidates to receive benralizumab in the individualized access program approved by national health authorities.

Primary Objective: To describe the demographic and baseline characteristics in patients with severe eosinophilic asthma who participated in the individualized access program approved in Spain and received at least one dose of benralizumab.

Secondary Objectives: To describe clinical outcomes in severe eosinophilic asthma patients who received at least three doses of benralizumab in the individualized access program.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years)
* Diagnosis of severe eosinophilic asthma requiring stable treatment of high doses of inhaled corticosteroids and a long-acting agonist β2 ± additional asthma controller
* Received at least one dose of benralizumab during the individualized access program period (March-December of 2018)
* Informed consent signed

Exclusion Criteria:

* Patients enrolled in a clinical trial who received benralizumab during the same period of the individualized access program
* Refuse to sign the informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be all patients who received at least one dose of benralizumab in individualized access program approved by the AEMPS.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Age | Up to 32 weeks
  Age (years)
Sex | Up to 32 weeks
  Male, Female
Body Mass Index (BMI) | Up to 32 weeks
  Weight and height will be combined to report BMI in kg/m^2
Smoking status | Up to 32 weeks
  Current smoker, Ex-smoker, Never smoker
Age at onset of asthma diagnosis | Up to 32 weeks
  Age (years)
Comorbidities | Up to 32 weeks
  Multiple response (binomial): allergies, nasal polyposis, rhinitis, GERD, atopic dermatitis, condition related with chronic OCS use, other eosinophilic driven diseases
Severe exacerbations | Up to 32 weeks
  Severe exacerbations in past 12 months: number and severity
Emergency room (ER) visits | Up to 32 weeks
  Number of ER visits
Hospitalizations | Up to 32 weeks
  Number of hospitalizations
Unscheduled visits | Up to 32 weeks
  Number of unscheduled visits
ACT | Up to 32 weeks
  ACT questionnaire score
miniAQLQ | Up to 32 weeks
  miniAQLQ questionnaire score
Blood eosinophils | Up to 32 weeks
  Blood eosinophils count (cells/microL)

SECONDARY OUTCOMES:
Incidence of severe exacerbations | Up to 32 weeks
  The incidence rate for any severe exacerbations in each calendar year will be calculated as follows: the sum of any severe exacerbations in that year divided by the total duration of follow-up in the same calendar year.

CONTACTS AND LOCATIONS:
Locations (1):
- BIG PAC, Madrid, Spain

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00052&attachmentIdentifier=a17b7040-7d5b-4c79-b9cd-4bed00284f5e&fileName=CSR_Summary_-_ORBE-Study.pdf&versionIdentifier=